CLINICAL TRIAL: NCT03058523
Title: Flavour Programming: Fruit and Vegetable Format Palatability
Brief Title: Flavour Programming: Fruit and Vegetable Palatability
Acronym: FLAVOUR
Status: Completed | Type: Observational
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/RINH/6 - Flavour; 16/LO/2238 (Other: NHS Research Ethics Committee Reference); 2-045-16 (Other: NHS REC Protocol number)
Record Dates: First submitted 2017-01-10; First posted 2017-02-23 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Child Development
Keywords: Flavour; Infants; Taste; Pregnancy; Programming; Fruit; Vegetables; Bitter profile; Food preferences
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tongue and cheek cells from buccal swabs
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Non-Pregnant: 30 non-pregnant women of childbearing age
- Pregnant: 30 pregnant women

SUMMARY:
Infants have an inborn preference for sweet and umami flavours and dislike sour and bitter, but there is evidence that sensory experiences beginning early in development can modify these preferences in favour ultimately of healthier food choices. Babies are first exposed to flavour in utero and then later through breast/formula milk. This can be manipulated to influence liking and consumption of individual foods with specific high-intensity flavours postnatally. There are no prospective studies evaluating the impact of increasing maternal fruit and vegetable intake during late pregnancy on a child's subsequent acceptance of fruit and vegetables, particularly those with a sour/bitter taste. The hypothesis is that an intervention to increase maternal intake of fruit and vegetables in late pregnancy will enhance fetal flavour exposure and make infants more likely to accept a wide variety of fruit and vegetables in childhood. Before testing this hypothesis, the investigators need to evaluate the general acceptance and taste profile of the fruit and vegetable formats that we intend to offer to pregnant women.

DETAILED DESCRIPTION:
Foods that tend to be rejected by children include those with the greatest importance for later health such as fruit and vegetables. Eating behaviour and acceptance of new tastes, textures and flavours in young children is influenced by a plethora of biological and environmental factors. Infants have an inborn preference for sweet and umami flavours and dislike sour and bitter, but there is evidence that sensory experiences beginning very early in development can positively modify these preferences in favour ultimately of healthier food choices. Babies are first exposed to flavour through swallowing amniotic fluid in utero and then later through breast or formula milk. There is evidence in a variety of species, including humans, to show that this can be manipulated particularly during late pregnancy to influence subsequent liking and consumption of individual foods with specific high intensity flavours potentially. However, there is a lack of prospective studies evaluating the impact of increasing maternal fruit and vegetable intake during late pregnancy on a child's subsequent acceptance of fruit and vegetables, particularly those with a bitter taste. The hypothesis is that an intervention to increase maternal intake of fruit and vegetables in late pregnancy, in women who normally struggle to achieve their 5-a-day, will enhance fetal flavour exposure and make infants more likely to accept a wide variety of fruit and vegetables in childhood. Before testing this hypothesis and designing the main study, investigators need to ensure that the component parts are feasible: central to this is evaluating the general acceptance and taste profile of the fruit and vegetable (F&V) formats that it is intended to offer to the mothers.

A range of innovative presentation formats for a variety of the most pungent fruits and vegetables are currently being developed. These include soups, sauces, crispbreads, muffins and smoothies that incorporate vegetables and/or fruits that are generally considered as bitter or sour tasting. A recent scoping survey of women of childbearing age confirmed prior observations in both sexes that vegetables with a bitter profile are less preferred / more likely never to have been tried, compared with sweet varieties. The survey also revealed that vegetables were largely consumed cooked and as part of ain meals. Accordingly the F&V formats to be evaluated are predominantly pre-cooked and designed to be warmed through in a microwave to avoid destruction and or leaching of flavour by over zealous cooking. Although the survey revealed low consumption of vegetables in smoothie form or as snacks, this may have been due to lack of easy availability and hence a number of these have been included to potentially increase diversity of dietary formats and flavour exposure.

This application is primarily a palatability trial to establish taste profile and general acceptability of the diverse F&V presentation formats in two groups: non-pregnant women of childbearing age, followed by pregnant women. As the perception of taste (particularly bitter, sweet and umami) may vary between individuals depending on genetic variation in certain taste receptor genes, it is proposed to characterise the relevant genotypes in buccal samples and relate this to their habitual diet and F&V preferences. The utility of a non-invasive sampling route for measuring expression of genes involved in taste perception will also be determined using tongue swabs as this is a desirable feature for potentially scrutinising any impact of the proposed intervention on the taste perception of mothers and their infants and also requires to be assessed ahead of the designing of the main intervention study.

ELIGIBILITY:
Inclusion Criteria:

* For the non-pregnant cohort: women of childbearing age with no major health issues and who currently struggle to meet the recommended 5 portions of fruit and vegetables per day.
* For the pregnant cohort: women who are >16 and <32 weeks pregnant (with no major health issues) and who currently struggle to meet the recommended 5 portions of fruit and vegetables per day.

Exclusion Criteria:

* Men and anyone who is unable to understand the participant information sheet and/or to speak, read or understand the English language (as the investigators do not have the resources to translate the materials)
* Women with known food allergies/intolerances or who are smokers, vegetarians or vegans
* Anyone using medication known to impact taste perception e.g. asthma inhalers
* Anyone with a hormone imbalance or metabolic disease that impacts their ability to taste
* Anyone with a history of an eating disorder
* Pregnant women with a history of recurring miscarriage or a diagnosis of hyperemesis gravidarium (severe nausea and vomiting), gestational diabetes or gestational hypertension or any other major pregnancy complication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women of Child bearing age
Sampling Method: Non-Probability Sample
Enrollment: 59 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Palatability of defined foods using a nine point scale | 9 months
  The two taste sessions will be done between 1 and 10 days apart dependant on volunteer availability

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Wallace, PhD, DSc, Principal Investigator — University of Aberdeen, The Rowett Institute, United Kingdom, AB25 2ZD
Locations (1):
- University of Aberdeen, The Rowett Institute, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: No